CLINICAL TRIAL: NCT05451264
Title: Study of the Effect of Hydrocortisone Administered for the Prevention of Pulmonary Bronchodysplasia (PREMILOC Trial) on the Determinants of Systemic Blood Pressure in Children
Brief Title: Study of the Effect of Hydrocortisone Administered for the Prevention of Pulmonary Bronchodysplasia (PREMILOC Trial) on the Determinants of Systemic Blood Pressure in Children (PREMILOCAP)
Acronym: PREMILOCAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: APHP211326
Record Dates: First submitted 2022-06-17; First posted 2022-07-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Infant, Premature, Diseases
MeSH Terms: conditions — Infant, Premature, Diseases | interventions — Blood Pressure Determination

STUDY DESIGN:
Intervention Model Description: Descriptive cross-sectional study of the subjects included in the double-blind, monocentric randomized controlled trial (children included and followed up at the Robert Debré hospital in the PREMILOC trial): follow-up of these children approximately 10 years later on vascular parameters
Who Masked: Participant, Care Provider, Investigator
Masking Description: The treatment having been received previously in the PREMILOC trial, no one knows which treatment the patients received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrocortisone (Experimental): During the PREMILOC trial, patients received hydrocortisone (0.5mg/kg/12h for 7 days and 0.5mg/kg/24h for 3 days).
  Interventions: Diagnostic Test: blood pressure measurement
- Placebo (Placebo Comparator): During the PREMILOC trial, patients received placebo (0.5mg/kg/12h for 7 days and 0.5mg/kg/24h for 3 days).
  Interventions: Diagnostic Test: blood pressure measurement

INTERVENTIONS:
Diagnostic Test: blood pressure measurement — Completion of the physical activity and quality of life questionnaire (PedSQL adapted to the age of the child), measurement of weight and height; Measurement of VOP (Pulse wave velocity), AI (increase index) and ECG (electro cardiogram) collection at rest lying down; Stimulation test by slow breathing at 6 cycles/min for three minutes; Continuation of the measurements in a standing position for 5 minutes; Installation of blood pressure holter (MAPA) which will be kept for 24 hours and then returned by post.

SUMMARY:
The risk of Arterial Hypertension (HTA) is increased in very premature infants and hydrocortisone administered in the neonatal period could modify this risk.

The main objective is to assess whether the administration of hydrocortisone in the perinatal period in children born prematurely is associated with an increase in Pulse Wave Velocity (PWV) by comparing the future of children included in the PREMILOC trial (hydrocortisone versus placebo) at the age of 7-13 years. The primary endpoint will be the carotid-femoral pulse wave velocity in m/s.

DETAILED DESCRIPTION:
Descriptive cross-sectional study of the subjects included in the double-blind, monocentric randomized controlled trial (children included and followed up at the Robert Debré hospital in the PREMILOC trial): follow-up of these children approximately 10 years later on vascular parameters.

ELIGIBILITY:
Inclusion Criteria:

* Child included in the PREMILOC trial on the Robert Debré site
* Age from 7 to 13 years old (eve of 14 years old)
* Consent of the holders of parental authority and agreement of the child

Exclusion Criteria:

* Absence of affiliation to a social security scheme
* Patient under state medical aid

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Velocity of the carotid-femoral pulse wave in m/s (VOP) | Inclusion
  Velocity of the carotid-femoral pulse wave in m/s measured by the SphygmoCor device.

SECONDARY OUTCOMES:
Index increase of VOP | Inclusion
  Index increase measured by the SphygmoCor device
Cardio-Radial Pulse Wave Velocity | Inclusion
  Cardio-Radial Pulse Wave Velocity in m/s (Biopac device); 3 measures: supine, standing and deep breaths
Sensitivity of the baroreflex | Inclusion
  Sensitivity of the baroreflex (up and down measurement, average; standing versus lying down: Biopac device) in ms/mmHg; 3 measures: supine, standing and deep breaths
High Frequence bare of the sympatho-vagal balance | Inclusion
  in ms^2; 3 measures: supine, standing and deep breaths
High Frequence bare of the sympatho-vagal balance | Inclusion
  in percent; 3 measures: supine, standing and deep breaths
Low frequence bare of the sympatho-vagal balance | Inclusion
  in percent; 3 measures: supine, standing and deep breaths
Low frequence bare of the sympatho-vagal balance | Inclusion
  in ms^2; 3 measures: supine, standing and deep breaths
Low Frequence/High Frequence ratio of the sympatho-vagal balance | Inclusion
  Low Frequence/High Frequence ratio of the sympatho-vagal balance
Parameters from ambulatory blood pressure measurement (ABPM) | During 24 hours
  Parameters from ambulatory blood pressure measurement (ABPM) (Spacelabs device) 24-hour systolic and diastolic average, day, night, systolic and diastolic nocturnal dipping
Other factors associated with the risk of early hypertension: quality of life | Data retrieved on inclusion
  quality of life: PedsQL quizz
Other factors associated with the risk of early hypertension: presence of overweight | Data retrieved on inclusion
  presence of overweight (yes/no)
Other factors associated with the risk of early hypertension: etnicity | Data retrieved on inclusion
  ethnicity
Other factors associated with the risk of early hypertension: daily physical activity | Data retrieved on inclusion
  daily physical activity: number of hours of physical activity per day
Other factors associated with the risk of early hypertension: Fetal growth restriction | Data retrieved on inclusion
  Fetal growth restriction during the pregnancy (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Chérine Chérine, MD PhD, Principal Investigator — APHP
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benzouid C, Bokov P, Coste P, Azonaha S, Diallo K, Guilmin-Crepon S, Baud O, Biran V, Delclaux C. Hydrocortisone administration in preterm infants is not associated with adverse cardiovascular outcomes in childhood. Pediatr Res. 2026 Jan 9. doi: 10.1038/s41390-025-04732-4. Online ahead of print. PMID 41513980